CLINICAL TRIAL: NCT00572988
Title: Symptom Management Intervention in Elderly CABG Patients
Brief Title: Symptom Management Intervention in Elderly Coronary Artery Bypass Patients
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0528-01-FB; R01NR007759 (NIH)
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Coronary Artery Disease
Keywords: symptom management; function status; physical activity; health care utilization
MeSH Terms: conditions — Coronary Artery Disease; Motor Activity; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The major purpose of this experimental study is to test the effects of the symptom management home care nursing intervention (SMHCNI) on recovery outcomes of elderly CABG patients, using a randomized, two group (n=284) repeated measures design with measurements at discharge, at 3 and 6 weeks, and 3 and 6 months postoperatively. One group will receive the intervention and routine care (RC) and the other group will receive RC only. The major aim will be to determine if the intervention group will demonstrate: better physiological functioning (decreased symptom interference on physical functioning; better scores on the SF36 subscales: physical, role-physical and vitality, and increased activity and exercise energy expenditure); better psychosocial functioning (decreased symptom interference on enjoyment of life; and better SF36 subscales; role-emotional, social, mental, and vitality); and fewer postoperative problems (e.g. infections, fluid in lungs, heart rate rhythm problems). Additional outcomes for secondary aims are: lower levels of health care utilization (HCU) (i.e., fewer number of visits to health care providers, fewer number of emergency department visits, fewer number of home health visits, fewer rehospitalizations); and higher patient satisfaction (with level of functioning and care received). In addition this study will examine the potential effects of mediating (evaluation of symptoms, and perceived self-efficacy), and moderating variables (participation in cardiac rehabilitation) with the intervention on outcomes identified.

DETAILED DESCRIPTION:
Effective follow-up and management of elderly post-CABG patients is important in the overall recovery process. Specifically, this study will attempt to bridge the gap in current literature related to the impact of follow-up interventions to enhance recovery outcomes in the CABG population. The major purpose of this experimental study is to test the effects of the symptom management home care nursing intervention (SMHCNI) on recovery outcomes of elderly CABG patients using a randomized, two group (N=284) repeated measures design with measurements at discharge, at 3 and 6 weeks, and 3 and 6 months post- operatively. One group will receive the intervention and routine care (RC) and the other group will receive only RC. The major aim will be to determine if the intervention group will demonstrate: better physiological functioning (decreased symptom interference on physical functioning (decreased symptom interference on physical functioning; better scores on the SF 36 subscales: physical, role-physical and vitality, and increased activity and exercise energy expenditure); better physiological conditioning (decreased symptom interference on physical functioning; better scores on the SF 36 subscales; role-emotional, social, mental, and vitality); and fewer post-operative problems (e.g., infections, fluid in lungs, heart rate rhythm problems). Additional outcomes for secondary aims are: lower levels of health care utilization [HCU] (i.e., fewer number of visits to health care providers, fewer number of emergency department visits, fewer number of home health visits, fewer rehospitalizations); and higher patient satisfaction (with level of functioning and care received). In addition this study will examine the potential effects of mediating (evaluation of level of functioning and care received)> In addition this study will examine the potential effects of mediating (evaluation of level of functioning and care received). In addition this study will examine the potential effects of mediating (evaluation of symptoms, and perceived self-efficacy, and moderating variables (participation in cardiac rehabilitation) with the intervention on outcomes identified above. The intervention will be delivered using a device called the Health Buddy that is attached to the patient's telephone line, able to download to a free secure Internet site daily, and cannot be used by health care providers for post-hospital follow up care. The 6- week SMHCNI was designed using Bandura's (1986) definition of self- efficacy which is to enhance the beliefs in ones capabilities to organize and execute the sources and actions required to manage prospective situations. Preliminary data have shown that these patients are going home with symptom management problems, but that complications arising from these problems might be prevented with early detection and management. Using a follow-up intervention such as the SMHCNI is expected to result in better functioning, management of symptoms and fewer post-operative problems. Also, a better understanding of HCU, patient satisfaction, and self-efficacy as variables will be described.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older and having undergone CABG surgery
* Oriented to person, place, and time
* Not visually impaired, able to hear, and able to speak and read English (eyeglasses and or hearing aids permitted)
* Not eligible for home health care (would not be homebound or have a draining wound)
* Have a phone with a non-rotary phone service
* Discharged within 7 days after surgery
* No physical impairments that would limit their physical functioning after surgery (e.g. stroke).

Exclusion Criteria:

* None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All subjects 65 and older who are admitted for a first time CABG surgery.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2002-05-01 (Actual); Study Completion 2007-01-01 (Actual)

PRIMARY OUTCOMES:
Symptom Evaluation | The duration of the study

SECONDARY OUTCOMES:
Functional Status | Duration of the study
Physical ACtivity | Duration of the Study
Health Care Utilization | 6 month follow up time period

CONTACTS AND LOCATIONS:
Overall Officials: Lani M Zimmerman, PhD, Principal Investigator — University of Nebraska